CLINICAL TRIAL: NCT04209829
Title: Response to Chimeric Antigen Receptor (CAR)-T Cells Therapy in Patients With Hematologic Malignancies (Lymphoma, Acute Lymphoblastic Leukemia, Multiple Myeloma) Depending on Tumor Characteristics
Brief Title: Response to Chimeric Antigen Receptor (CAR)-T Cells Therapy in Patients With Hematologic Malignancies Depending on Tumor Characteristics
Acronym: BIOCART-HM
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190678
Record Dates: First submitted 2019-11-22; First posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-10

CONDITIONS: Hematologic Diseases
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with haematological malignancy: Patients, aged 15 years or over, with haematological malignancy (Lymphoma, ALL, MM) integrated into a CAR-T Cells program treatment

SUMMARY:
Immunotherapy with Chimeric Antigen Receptor (CAR) T Cells, T cells whose receptor has been genetically modified, is based on improving the immune response against the tumor. This approach is promising for patients with hematologic malignancies refractory to chemotherapy. Despite impressive results, too many patients are relapsing. The reasons for the relapse, after the injection of CAR T cells, need to be explored. In this context of newly introduced therapeutics, it is essential to better understand the factors associated with the response to treatment with CAR T Cells, especially the characteristics of the tumor and its microenvironment.

The objective of this study is to understand the role of tumor biology, and its microenvironment, in the response to CAR-T Cells therapy in patients with hematologic malignancies

ELIGIBILITY:
Inclusion Criteria:

* patient with hematological malignancy (lymphoma, ALL, MM)
* patient integrated into a CAR-T Cells program treatment
* patient aged 15 years or over
* patient having signed a written consent; as well as his legal representative if <18 years old

Exclusion Criteria:

* patient with other hematological malignancies than lymphoma, LAL or MM
* patient's weight <58 kg
* patient treated with another treatment than CAR-T Cells
* patient under tutorship or curatorship
* patient not covered by a health system

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hematological malignancy
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2035-03 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | 90 days after (CAR)-T cell therapy initiation

SECONDARY OUTCOMES:
Overall Survival rate | 1 year
Objective response rate | 30 days
Objective response rate | 90 days
Objective response rate | 1 year
Objective response rate | 2 years
Objective response rate | 5 years
Objective response rate | 10 years
Progression-free survival | at 1 year
Incidence of adverse events | at 30 days
Incidence of adverse events | at 90 days
Incidence of adverse events | at 1 year
Incidence of adverse events | at 2 years
Incidence of adverse events | at 5 years
Incidence of adverse events | at 10 years
Proportion of patients with an admission in intensive care | at 30 days
Proportion of patients with an admission in intensive care | at 90 days
Severity of neurological toxicities | at 30 days
  Severity of neurological toxicities will be assessed by physical, and by Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Severity of neurological toxicities | at 90 days
  Severity of neurological toxicities will be assessed by physical examination and by Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Severity of neurological toxicities | at 6 months
  Severity of neurological toxicities will be assessed by physical, cognitive examination and by Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Severity of neurological toxicities | at 2 years
  Severity of neurological toxicities will be assessed by physical examination and by Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Severity of neurological toxicities | at 5 years
  Severity of neurological toxicities will be assessed by physical examination and by Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Severity of neurological toxicities | at 10 years
  Severity of neurological toxicities will be assessed by physical examination and by Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Proportion of patients with a cytokine release syndrome | at baseline
  Cytokine release syndrome will be assessed by CTCAE v5.0
Proportion of patients with a cytokine release syndrome | at 7 days
  Cytokine release syndrome will be assessed by CTCAE v5.0
Proportion of patients with a cytokine release syndrome | at 30 days
  Cytokine release syndrome will be assessed by CTCAE v5.0

IPD SHARING:
Plan to Share IPD: Undecided